CLINICAL TRIAL: NCT00547625
Title: A Multicenter, Parallel-Arm, Placebo-Controlled, Double-Blind Study to Evaluate the Efficacy and Safety of Tadalafil Administered Once Daily to Men With Lower Urinary Tract Symptoms Secondary to Benign Prostatic Hyperplasia
Brief Title: Study to Determine Safety and Effectiveness of Tadalafil on Prostate Related Sex Organ/Urinary Tract Problems
Acronym: PILUTS
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Eli Lilly and Company (Industry)
Collaborators: ICOS Corporation (Industry)
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: 9120; H6D-MC-LVGC
Record Dates: First submitted 2007-10-18; First posted 2007-10-22 (Estimated); Last update posted 2007-10-22 (Estimated); Status verified 2007-10

CONDITIONS: Prostatic Hyperplasia; Prostate
MeSH Terms: conditions — Prostatic Hyperplasia | interventions — Tadalafil

STUDY DESIGN:
Who Masked: Participant, Investigator
Oversight: Data Monitoring Committee: No

ARMS (2):
- 1 (Placebo Comparator): Placebo run in followed by 5 mg treatment phase 1 and then 20 mg treatment phase 2 which both include a placebo control.
  Interventions: Drug: placebo
- 2 (Active Comparator): Treatment phase 1 includes 5 mg tadalafil 6 weeks then treatment phase 2 which includes 20 mg tadalafil for 6 weeks.
  Interventions: Drug: tadalafil

INTERVENTIONS:
Drug: tadalafil — Treatment phase 1 includes 5 mg tadalafil tablet taken by mouth once a day for 6 weeks then treatment phase 2 which includes 20 mg tadalafil tablet taken by mouth once a day for 6 weeks.
  Other Names: LY450190; Cialis; IC351
  Arms: 2
Drug: placebo — Placebo tablet run in followed by placebo treatment period with one tablet taken by mouth once a day for twelve weeks.
  Arms: 1

SUMMARY:
Study to look at safety and effectiveness of different doses of tadalafil on prostate related genital/urinary tract problems.

ELIGIBILITY:
Inclusion Criteria:

* 6 month history of lower urinary tract symptoms either obstructive and/or irritative secondary to prostate related problems as diagnosed by a urologist.
* Stopped using treatments at least four weeks prior to study and agree to not use any other treatments during the study.
* Meet required prostate symptom score and urine flow rate.

Exclusion Criteria:

* Serum prostate specific antigen (PSA) greater than 10 (between 4 and 10, inclusive, without a negative biopsy w/in the last 6 months.
* Prostate removal and various other pelvic surgeries.
* Neurological disease or condition known to affect the bladder.
* Clinical evidence of prostate cancer, urinary tract inflammation or infection, including prostatitis.
* Have taken medications such as nitrates, finasteride, or dutasteride within the year.

Min Age: 45 Years | Sex: Male | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 275 (Actual)
Dates: Start 2004-10; Study Completion 2005-07 (Actual)

PRIMARY OUTCOMES:
International Prostate Symptom Score (IPSS) sum total of questions 1-7 | 6 and 12 weeks

SECONDARY OUTCOMES:
Evaluate different domains of the IPSS sums along with other questionnaires such as the LUTS GAQ and BII. | 12 weeks
Measure Uroflowmetry parameters | 12 weeks
Evaluate safety by PSA levels and postvoid residual volume (PVR) | 12 weeks

CONTACTS AND LOCATIONS:
Overall Officials: Call 1-877-CTLILLY (1-877-285-4559) or 1-317-615-4559 Mon - Fri 9 AM - 5 PM Eastern time (UTC/GMT - 5 hours, EST), Study Director — Eli Lilly and Company
Locations (1):
- For additional information regarding investigative sites for this trial, contact 1-877-CTLILLY (1-877-285-4559, 1-317-615-4559) Mon- Fri from 9 AM to 5 PM Eastern Time (UTC/GMT - 5 hours, EST), or speak with your personal physician., Chicago, Illinois, United States

REFERENCES:
- See also: Lilly Clinical Trial Registry — http://www.lillytrials.com